CLINICAL TRIAL: NCT04847531
Title: REVEAL-CKD: A Retrospective, Multinational Observational Study to Determine the Prevalence and Consequences of Undiagnosed Chronic Kidney Disease
Brief Title: REVEAL-CKD: Prevalence and Consequences of Undiagnosed Chronic Kidney Disease
Acronym: REVEAL-CKD
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D169AR00003
Record Dates: First submitted 2021-03-29; First posted 2021-04-19 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2024-12

CONDITIONS: Chronic Kidney Disease
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Stage 3 chronic kidney disease patients: Patients with two consecutive eGFR measurements indicating stage 3 CKD (≥30 and <60 mL/min/1.73m2) during the observation period

SUMMARY:
This is a retrospective, multinational, non-interventional, observational study. A series of cohort studies will be conducted to assess the prevalence of undiagnosed stage 3 CKD in each region. The study will also assess the current state of CKD management in patients with undiagnosed CKD

DETAILED DESCRIPTION:
This study is a retrospective, multinational, non-interventional observational study. The study does not attempt to test any specific a priori hypothesis; it is descriptive only and will collect data under conditions of routine medical care. Relevant secondary databases will be identified, and a series of cohort studies will be conducted to assess the prevalence of undiagnosed CKD. The study will also assess the current state of CKD management in patients with undiagnosed CKD.

Primary Objectives

1. Estimate the point prevalence of undiagnosed stage 3 CKD (proportion of patients with eGFR measurements indicating stage 3 CKD with no corresponding CKD diagnostic code either before or up to six months after the second abnormal eGFR value)
2. Describe time to CKD diagnosis in patients with no prior CKD diagnosis code at index date (time of second qualifying eGFR), overall and by patient characteristics

Secondary Objectives

1. Assess trends in the prevalence (point prevalence) of undiagnosed CKD by calendar year
2. Describe baseline characteristics among those with undiagnosed versus diagnosed CKD
3. Assess CKD management and monitoring practices (post index date) in patients with diagnosed versus undiagnosed CKD

Exploratory objectives (pending feasibility)

1. Describe the risk of selected adverse clinical outcomes longitudinally among those with undiagnosed versus diagnosed CKD
2. Describe HCRU associated with undiagnosed versus diagnosed CKD
3. Assess association between the timing of the CKD diagnosis and the risk of selected adverse clinical outcomes and HCRU in patients with no CKD diagnosis code prior to the index date
4. Describe health care costs associated with undiagnosed versus diagnosed CKD
5. For CKD patients with eGFR 25-75 mL/min/1.73m2 and urine albumin creatinine ratio (UACR) 200 - 5000 mg/g (DAPA-CKD trial-like population):

   1. Estimate the point prevalence of undiagnosed CKD
   2. Describe the risk of selected adverse clinical outcomes longitudinally among those with undiagnosed CKD
   3. Describe HCRU and costs associated with undiagnosed CKD

ELIGIBILITY:
Inclusion Criteria:

* At least two consecutive eGFR laboratory tests with values ≥30 and <60 mL/min/1.73 m2 (Stage 3A or 3B) that are >90 and ≤730 days apart. The index date is the date of the second eGFR measure meeting the criteria for stage 3 CKD
* At least 12 months of continuous presence in the database or registration in the data prior to the first qualifying eGFR (for data sources with information on enrolment)
* Age ≥18 years at index date

Exclusion Criteria:

* Solid organ transplant before the study index date
* Any evidence of advanced CKD (stage 4, 5) based on CKD diagnostic codes, or renal replacement therapy before the index date

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients ≥18 years old with two consecutive eGFR measurements indicating stage 3 CKD (≥30 and <60 mL/min/1.73m2 using CKD-EPI (preferred) or MDRD equation) recorded more than 90 days apart (max. 730 days), meeting the inclusion criteria will be included in the study (from 2015 onwards).
Sampling Method: Non-Probability Sample
Enrollment: 1006361 (Actual)
Dates: Start 2020-12-15 (Actual); Primary Completion 2023-11-13 (Actual); Study Completion 2023-11-13 (Actual)

PRIMARY OUTCOMES:
Prevalence of undiagnosed stage 3 chronic kidney disease (CKD) | From 2015 assessed throughout the study, up to a maximum of 8 years
  Undiagnosed stage 3A-3B CKD identified as having no healthcare encounter with a diagnosis code for CKD any time before or up to six months post index date (date of second consecutive estimated glomerular filtration rate [eGFR] value indicating stage 3 CKD recorded at least 90 days after the first abnormal eGFR value), assessed overall and by calendar year
Time to CKD diagnosis | From second abnormal eGFR value until the date of CKD diagnosis or end of follow-up, assessed throughout the study period, up to a maximum of 5 years
  Time to CKD diagnosis in patients no CKD diagnosis code any time prior to laboratory measurements indicating stage 3 CKD

SECONDARY OUTCOMES:
Describe proportion of patients comorbidities and other patient characteristics | From 2015 assessed throughout the study, up to a maximum of 8 years
  Describe patient characteristics including demographics, clinical assessments, family history, procedures, laboratory measurements, treatment patterns and clinical history (comorbidities) stratified by CKD diagnosis status
Proportion of patients monitored for kidney function and complications | From six months after the second abnormal eGFR measurement, assessed throughout the study period until end of follow-up, up to a maximum 18 months
  * Serum Cr test (outpatient)
  * Patients receiving a UACR test (outpatient)
  * Serum calcium
  * Phosphate
  * Albumin
  * Bicarbonate
  * Potassium
  * Hemoglobin
  * Albuminuria
Proportion of patients tested for CKD | From six months after the second abnormal eGFR measurement, assessed throughout the study period until end of follow-up, up to a maximum 6 months
  - UACR test
Proportion of patients prescribed selected medications | From six months after the second abnormal eGFR measurement, assessed throughout the study period until the end of follow-up, up to a maximum 5 years
  * Statin prescription
  * Angiotensin converting enzyme inhibitors (ACEis) or angiotensin receptor blockers (ARBs)
  * Sodium-glucose cotransporter-2 (SGLT2) inhibitors
  * Vaccination (influenza)
Proportion of patients monitored for high blood pressure | From six months after the second abnormal eGFR measurement, assessed throughout the study period until end of follow-up, up to a maximum 5 years
  * Patients receiving BP measurement
  * BP measurement ≤140/90
  * BP measurement ≤ 130/80 in patients with evidence of albuminuria and/or diabetes
Proportion of patients monitored for glycaemic control | From six months after the second abnormal eGFR measurement, assessed throughout the study period until end of follow-up, up to a maximum 5 years
  - HbA1c test in patients with diabetes
Proportion of patients receiving kidney function monitoring after initiation of angiotensin receptor blocker or angiotensin converting enzyme inhibitors | From six months after the second abnormal eGFR measurement, assessed throughout the study period until end of follow-up, up to a maximum 5 years
  - An outpatient serum creatinine measurement

OTHER OUTCOMES:
Incidence of adverse renal events | From six months after the second abnormal eGFR until the date of an adverse renal outcome, assessed throughout the study until end of follow-up, up to a maximum of 5 years
  * Sustained ≥50% reduction in eGFR; or
  * End stage kidney disease (ESKD); defined as a composite of chronic dialysis, renal transplant, or sustained eGFR<15mL/min/1.732 (at least two consecutive measures ≥28 days apart)
Incidence of all-cause mortality | From six months after the second abnormal eGFR until death due to any cause, assessed throughout the study until end of follow-up, up to a maximum of 5 years
  All-cause mortality
CKD progression | From six months after the second abnormal eGFR until the date of CKD progression, assessed throughout the study until end of follow-up, up to a maximum of 5 years
  Progression to CKD stage 4 or higher
Incidence of Cardiovascular (CV) events | From six months after the second abnormal eGFR until the date of a CV event, assessed throughout the study until end of follow-up, up to a maximum of 5 years
  * Composite of non-fatal MI, non-fatal stroke, or CV death
  * Composite of non-fatal MI, non-fatal stroke, or all-cause mortality)
  * Composite of non-fatal MI, non-fatal stroke, hospitalization for unstable angina, hospitalization for heart failure, or CV death
  * Stroke
  * Hospitalisation for heart failure
Describe health care resource utilisation and associated costs | From six months after the second abnormal eGFR, assessed throughout the study until end of follow-up, up to a maximum of 5 years
  To understand the healthcare resource use and cost associated with undiagnosed CKD

CONTACTS AND LOCATIONS:
Overall Officials: Navdeep Tangri, Principal Investigator — University of Manitoba
Locations (13):
- United States (3):
  - Research Site, Louisville, Kentucky
  - Research Site, Cambridge, Massachusetts
  - Research Site, Ann Arbor, Michigan
- Research Site, Sydney, New South Wales, Australia
- Research Site, São Paulo, Brazil
- Research Site, Kingston, Ontario, Canada
- Research Site, Guangzhou, Guangdong, China
- Research Site, Boulogne-Billancourt, France
- Research Site, Frankfurt, Germany
- Research Site, Milan, Italy
- Research Site, Kyoto, Japan
- Research Site, Madrid, Spain
- Research Site, London, Greater London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the deidentified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- [Derived] Tangri N, Moriyama T, Schneider MP, Virgitti JB, De Nicola L, Arnold M, Barone S, Peach E, Wittbrodt E, Chen H, Jarbrink K, Kushner P. Prevalence of undiagnosed stage 3 chronic kidney disease in France, Germany, Italy, Japan and the USA: results from the multinational observational REVEAL-CKD study. BMJ Open. 2023 May 22;13(5):e067386. doi: 10.1136/bmjopen-2022-067386. PMID 37217263
- [Derived] Tangri N, Peach EJ, Franzen S, Barone S, Kushner PR. Patient Management and Clinical Outcomes Associated with a Recorded Diagnosis of Stage 3 Chronic Kidney Disease: The REVEAL-CKD Study. Adv Ther. 2023 Jun;40(6):2869-2885. doi: 10.1007/s12325-023-02482-5. Epub 2023 May 3. PMID 37133647
- See also: The CSR synopsis_D169AR00003 — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D169AR00003&attachmentIdentifier=562af12c-16b4-4aeb-afa2-ceeee0ccaf80&fileName=REVEAL_CKD_study_report_synopsis_D169AR00003.pdf&versionIdentifier=